CLINICAL TRIAL: NCT01430754
Title: A Randomized Withdrawal Study to Demonstrate the Maintenance of Effect of 20 mg Tasimelteon in the Treatment of N24HSWD
Brief Title: Withdrawal Study to Demonstrate the Maintenance Effect in the Treatment of Non-24-Hour Sleep-Wake Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VEC-162-3203
Record Dates: First submitted 2011-08-30; First posted 2011-09-08 (Estimated); Results first posted 2014-10-10 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Non-24-Hour Sleep-Wake Disorder
Keywords: Blindness; Eye Diseases; Nap Disorders; Circadian Rhythm Disorders; Sleep Disorders; Circadian Rhythm Sleep Disorders; Dyssomnias; Nervous System Diseases
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Blindness; Eye Diseases; Chronobiology Disorders; Sleep Wake Disorders; Dyssomnias; Nervous System Diseases | interventions — tasimelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tasimelteon (Experimental): 20 mg tasimelteon capsules
  Interventions: Drug: tasimelteon
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tasimelteon — 20 mg tasimelteon capsules, daily
  Other Names: VEC-162
  Arms: tasimelteon
Drug: Placebo — Placebo capsules, daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the maintenance effect and safety of 20 mg tasimelteon versus placebo in subjects suffering from Non-24-Hour Sleep-Wake Disorder.

DETAILED DESCRIPTION:
Non-24-Hour Sleep-Wake Disorder (N24HSWD) occurs when individuals are unable to synchronize their endogenous circadian pacemaker to the 24-hour light-dark cycle, and the timing of their circadian rhythm instead reflects the intrinsic period of their endogenous circadian pacemaker. As a result, the circadian rhythm of sleep-wake propensity in these individuals moves gradually later and later each day if there circadian period is > 24 hours and earlier and earlier is < 24 hours. These individuals will be able to sleep well at night when their sleep-wake propensity rhythm is approximately aligned with the 24-hour light-dark and social cycle. However, after a short time, the endogenous sleep-wake propensity rhythm and the 24-hour light-dark cycle will move out of synchrony with each other, and they may have difficulty falling asleep until well into the night. In addition to problems sleeping at the desired time, the subjects experience daytime sleepiness and daytime napping. As time progresses, the endogenous circadian rhythm of sleep-wake propensity in these individuals moves further and further away from the 24-hour light-dark cycle and gradually, these individuals are unable to sleep at night and as a result experience extreme sleepiness during the daytime hours and more frequent naps with a longer duration. Eventually, the sleep-wake time moves back into alignment with the social time for sleep and the individuals sleep well at night and have decreased daytime napping. The alignment between their endogenous circadian rhythms and the 24-hour day is temporary as they are continually drifting later and later each day.

This will be a multicenter, randomized withdrawal, double-masked, placebo-controlled, parallel study. The study has three phases: the tasimelteon run-in phase, the tau estimation phase, and the randomized withdrawal phase. Subjects who have participated in study VP-VEC-162-3201 that meet the entry criteria for this study will be eligible for the run-in phase The run-in phase comprises a screening visit where subject's initial eligibility will be evaluated. Subjects that meet the inclusion/exclusion criteria at screening will enter the run-in phase and will be dosed with 20 mg of tasimelteon daily for 6 weeks. The tau estimation phase (48 hour urine collection samples to evaluate response to tasimelteon) will follow the run-in phase and will last approximately 6 weeks long. The randomized withdrawal phase comprises approximately eight weeks of treatment with either placebo or tasimelteon 20 mg taken approximately 1 hour prior to their target bedtime in a double-masked fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and acceptance to provide informed consent;
2. Males, non-fecund females (i.e., surgically sterilized, if procedure was done 6 months before screening or subject is postmenopausal, without menses for 6 months before screening), or females of child-bearing potential using an acceptable method of birth control for a period of 35 days before the first dosing and must have a negative pregnancy test at the screening and baseline visits; Note: Women using hormonal methods of birth control must use an additional method of birth control during the study and for one month after the last dose.
3. Willing and able to comply with study requirements and restrictions including a commitment to a fixed 9-hour sleep opportunity during the study;
4. Diagnosis of N24HSWD in a previous clinical trial as measured by a tau value of > 24.1 and the lower bound of the 95% CI is > 24.

Exclusion Criteria:

1. History (within the 12 months prior to screening) of psychiatric disorders including Major Depressive Disorder, Generalized Anxiety Disorder, Axis II Disorders, delirium or any other psychiatric disorder, that is not being successfully treated or has not been resolved and that in the opinion of the clinical investigator would affect participation in the study or full compliance with study procedures;
2. History of intolerance and/or hypersensitivity to melatonin or melatonin agonists;
3. History of drug or alcohol abuse as defined in DSM-IV, Diagnostic Criteria for Drug and Alcohol Abuse, within the 12 months prior to screening and/or regular consumption of alcoholic drinks (> 2 drinks/day or > 14 drinks/week);

   a. Note: A standard drink is equal to 13.7 grams (0.6 ounces) of pure alcohol or
   * 12-ounces of beer
   * 8-ounces of malt liquor
   * 5-ounces of wine
   * 1.5-ounces or a "shot" of 80-proof distilled spirits or liquor (e.g., gin, rum, vodka, or whiskey);
4. Subject is at risk of suicide, in the opinion of the Investigator. Evidence of suicide risk could include any suicide attempt within the past year or any other suicidal behavior within the past year;
5. Current clinically significant cardiovascular, respiratory, neurologic, hepatic, hematopoietic, renal, gastrointestinal or metabolic dysfunction unless currently controlled and stable;
6. Subjects who have estimated creatinine clearance (CLcr; based on the Cockcroft-Gault equation) ≤ to 55 mL/min;
7. Clinically significant deviation from normal in clinical laboratory results, vital signs measurements, or physical examination findings at screening as determined by the clinical investigator;
8. Indication of impaired liver function (values for AST, ALT or bilirubin > 2 times Upper Limit of Normal);
9. Pregnant or lactating females;
10. A positive test for drugs of abuse at the screening visit; Note: A positive drug screen at Visit 1 needs to be discussed with the medical monitor and will be evaluated on a case-by-case basis.
11. Smoke more than 10 cigarettes/day;
12. Worked night, rotating, or split (period of work, followed by break, and then return to work) shift work within 1 month of the screening visit or plan to work these shifts during the study;
13. Unwilling or unable to follow the medication restrictions described in Section 8.2., or unwilling or unable to sufficiently wash-out from use of a restricted medication
14. Unable to perform calls to the study IVR system to report questionnaire results;
15. Any other sound medical reason as determined by the clinical investigator;
16. Legal incompetence or limited legal competence, detainment in an institution for official or legal reasons.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanda Pharmaceuticals, Study Director — Vanda Pharmaceuticals
Locations (22):
- United States (22):
  - Pulmonary Associates, PA, Phoenix, Arizona
  - SDS Clinical Trials Inc., Orange, California
  - VA Palo Alto Health Care System/PAIRE (San Fransisco Bay Area), Palo Alto, California
  - St. Johns Sleep Disorder Center - St. Johns Medical Plaza, Santa Monica, California
  - Radiant Research - Denver, Denver, Colorado
  - PAB Clinical Research Inc., Brandon, Florida
  - Kendall South Medical Center, Inc., Miami, Florida
  - Ocean Sleep Disorders Center - Ormond Beach, Ormond Beach, Florida
  - Sleep Disorders Center Of Georgia, Atlanta, Georgia
  - Suburban Lung Associates SC, Elk Grove Village, Illinois
  - The Center for Sleep and Wake Disorders (Washington, D.C. Metropolitan Area), Chevy Chase, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Michigan Head-Pain Neurological Institute, Ann Arbor, Michigan
  - St. Luke's Sleep Medicine and Research Center (St. Louis Metropolitan Area), Chesterfield, Missouri
  - New York Eye and Ear Infirmary, New York, New York
  - Ohio Sleep Medicine Institute (Columbus Metropolitan Area), Dublin, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Columbia Research Group Inc., Portland, Oregon
  - Mercy Fitzgerald Hospital - Sleep Disorders Center (Philadelphia Metropolitan Area), Lafayette Hill, Pennsylvania
  - Consolidated Clinical trials, Pittsburgh, Pennsylvania
  - SleepMed, Inc. - Columbia, Columbia, South Carolina
  - Todd J. Swick, M.D., P.A., Houston, Texas

REFERENCES:
- [Derived] Lockley SW, Dressman MA, Licamele L, Xiao C, Fisher DM, Flynn-Evans EE, Hull JT, Torres R, Lavedan C, Polymeropoulos MH. Tasimelteon for non-24-hour sleep-wake disorder in totally blind people (SET and RESET): two multicentre, randomised, double-masked, placebo-controlled phase 3 trials. Lancet. 2015 Oct 31;386(10005):1754-64. doi: 10.1016/S0140-6736(15)60031-9. Epub 2015 Aug 4. PMID 26466871

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who met the I/E criteria were treated with tasimelteon 20 mg for 6 wks during run-in. Entrained patients were randomized to tasimelteon 20 mg or placebo for the remainder of the study.
Period: Run-In Phase
Arm/Group | Tasimelteon | Placebo
Started | 57 | 0 (During the run-in phase, participants were treated with tasimelteon only.)
Entrained - After Run-In Phase | 24 | 0
Completed | 20 (Defined as the number of patients who entered the randomized-withdrawal phase) | 0
Not Completed | 37 | 0
Not completed — Circadian Period Ineligible | 24 | 0
Not completed — Protocol Violation | 6 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Other | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Randomized Phase
Arm/Group | Tasimelteon | Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Run-In - Not Randomized includes the demographics for patients who participated in the run-in phase but who were not randomized.
Groups:
- Run-In - Not Randomized: 20 mg tasimelteon capsules
  tasimelteon: 20 mg capsules, daily
- Tasimelteon (Randomized): 20 mg tasimelteon capsules
  tasimelteon: 20 mg tasimelteon capsules, daily
- Placebo (Randomized): Placebo capsules
  Placebo: Placebo capsules, daily
- Total: Total of all reporting groups
Arm/Group | Run-In - Not Randomized | Tasimelteon (Randomized) | Placebo (Randomized) | Total
Number analyzed (Participants) | 37 | 10 | 10 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (13.18) | 51.3 (12.87) | 52.1 (12.01) | 52.1 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 4 | 4 | 24
  Male | 21 | 6 | 6 | 33

OUTCOME MEASURES:

1. Primary Outcome: Maintenance of Entrainment (aMT6s) in Subjects With N24HSWD.
Description: Entrainment is a measure of synchronization of the master body clock to the 24-hour day. The circadian period (τ) was calculated using urinary aMT6s collected over four separate 48 hour periods, approximately 1 week apart, during the run-in and randomized phases of the trial. Maintenance of entrainment is defined as the proportion of subjects who become non-entrained to a 24 hour day after randomization to tasimelteon or placebo. Non-entrainment was defined as having a post-baseline τ value ≥ 24.1 or the lower bound of the 95% CI >24.0.
Time Frame: Approximately 12 weeks
Measure: Number; unit: participants
Arm/Group | Tasimelteon | Placebo
Number analyzed (Participants) | 10 | 10
participants | 9 | 2

2. Secondary Outcome: Maintenance of Entrainment (Cortisol) in Subjects With N24HSWD
Description: Entrainment is a measure of synchronization of the master body clock to the 24-hour day. The circadian period (τ) was calculated using urinary cortisol collected over four separate 48 hour periods, approximately 1 week apart, during the run-in and randomized phases of the trial. Maintenance of entrainment is defined as the proportion of subjects who become non-entrained to a 24 hour day after randomization to tasimelteon or placebo. Non-entrainment was defined as having a post-baseline τ value ≥ 24.1 or the lower bound of the 95% CI >24.0.
Time Frame: Approximately 12 weeks
Measure: Number; unit: participants
Arm/Group | Tasimelteon | Placebo
Number analyzed (Participants) | 10 | 10
participants | 8 | 2

3. Secondary Outcome: Change From Run-In in Subjective Nighttime Total Sleep Time in Lower Quartile of Days (LQ-nTST) During the Randomized Phase
Description: LQ-nTST measures the average nighttime sleep during the patient's worst 25% of nights (shortest total nighttime sleep) from run-in and randomized phase. The higher number indicates improvement.
Time Frame: Approximately 12 weeks
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Tasimelteon | Placebo
Number analyzed (Participants) | 10 | 10
minutes | -6.74 (18.986) | -73.74 (18.986)

4. Secondary Outcome: Change From Run-In in Total Daytime Sleep Duration in Lower Quartile of Days (UQ-dTSD) During the Randomized Phase
Description: UQ-dTSD measures the average daytime sleep during the patient's worst 25% of days (longest total daytime sleep) from run-in and randomized phase. Lower number indicates improvement.
Time Frame: Approximately 12 weeks
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Tasimelteon | Placebo
Number analyzed (Participants) | 10 | 10
minutes | -9.31 (17.253) | 49.95 (17.253)

5. Secondary Outcome: Change From Run-In in Midpoint of Sleep (MoST) During the Randomized Phase
Description: Midpoint of Sleep Timing (MoST) is the measurement of the average timing of sleep relative to bedtime. The average MoST value will trend to 0 as an individual's sleep becomes more fragmented. Improvement is defined as an increase in the average.
Time Frame: Approximately 12 weeks
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Tasimelteon | Placebo
Number analyzed (Participants) | 10 | 10
minutes | 19.99 (8.611) | -16.05 (8.611)

6. Secondary Outcome: Change From Run-In in Circadian Time to Relapse During the Randomized Phase
Description: Time to relapse is defined as a 45 minute or greater decrement in the weekly average of subjective nighttime total sleep time (nTST) compared to the Run-in Phase.
Time Frame: Approximately 8 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Tasimelteon | Placebo
Number analyzed (Participants) | 10 | 10
days | NA [NA to NA] — Circadian time to relapse never gets as low as 50% (median). | 24.7 [11.1 to 44.4]

ADVERSE EVENTS:
Time Frame: 1st dose to 30 days following last administration of study treatment
Groups:
- Total Run-In; Tasimelteon: 20 mg tasimelteon capsules
  tasimelteon: 20 mg tasimelteon capsules, daily
Arm/Group | Total Run-In | Run-In - Not Randomized | Tasimelteon | Placebo
Serious Adverse Events (participants affected / at risk) | 1/57 | 0/37 | 2/10 | 0/10
Other Adverse Events (participants affected / at risk) | 16/57 | 10/37 | 5/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Run-In (N=57) | Run-In - Not Randomized (N=37) | Tasimelteon (N=10) | Placebo (N=10)
Serotonin Syndrome (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Run-In (N=57) | Run-In - Not Randomized (N=37) | Tasimelteon (N=10) | Placebo (N=10)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Blood creatine phosphokinase (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Crystal urine present (Investigations) | 2 (3) | 2 (3) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (4) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 2 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No